CLINICAL TRIAL: NCT00865761
Title: A Relative Bioavailability Study of 3 mg Alprazolam Extended Release Tablets Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Alprazolam 3 mg ER Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R05-0851
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Alprazolam; Healthy subjects
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Alprazolam 3 mg Extended Release Tablets, single dose
  Interventions: Drug: Alprazolam 3 mg Extended Release Tablets, single dose
- B (Active Comparator): XANAX XR® 3 mg tablets, single dose
  Interventions: Drug: XANAX XR® 3 mg tablets, single dose

INTERVENTIONS:
Drug: Alprazolam 3 mg Extended Release Tablets, single dose — A: Experimental Subjects received Alpharma formulated products under fasting conditions
  Other Names: Alprazolam
  Arms: A
Drug: XANAX XR® 3 mg tablets, single dose — B: Active comparator Subjects received Pharmacia & Upjohn Company formulated products under fasting conditions
  Other Names: Alprazolam
  Arms: B

SUMMARY:
The purpose of this study is to compare the relative bioavailability of 3 mg Alprazolam Extended Release Tablets by Alpharma with that of 3 mg XANAX XR® Tablets by Pharmacia & Upjohn Company following a single oral dose (1 x 3 mg extended-release tablet) in healthy adult volunteers administrated under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, single-dose, two-way crossover study under fasting conditions.

Official Title: A Relative Bioavailability Study of 3 mg Alprazolam Extended Release Tablets Under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men and women 18 years of age or older at the time of dosing. The weight range will not exceed ± 20% for height and body frame as per Desirable Weights for Adults -1983 Metropolitan Height and Weight Table.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:

  * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential; RBC count, platelet count
  * CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
  * HIV antibody and hepatitis B surface antigen screens;
  * URINALYSIS: by dipstick, microscopic examination if dipstick positive; and.
  * URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
  * SERUM PREGNANCY SCREEN (female volunteers only)
  * FSH (to verify postmenopausal status; female volunteers only)
* If female and:

  * is postmenopausal for at least I year and has a serum FSH level ≥ 30 mIU/mL; or
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the medical investigator).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen, hepatitis C antibody or HIV antibody.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to alprazolam or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the medical investigator).
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic• drug metabolism in the 28 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing.
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson,, Pharm.D,, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States